CLINICAL TRIAL: NCT07097428
Title: Individualized Temperature Health Risk Early Warning for Reducing the Recurrence Risk of Stroke:A Multicenter, Randomized Controlled Trial Study
Brief Title: An Application Provides Temperature-related Health Risk Warnings and Protective Recommendations on Stroke
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: [2024]444-003-1-1
Record Dates: First submitted 2025-06-19; First posted 2025-07-31 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Temperature health risk early warning (Experimental): Receive individualized temperature health risk warning through the application
  Interventions: Other: Temperature health risk early warning
- Routine education (No Intervention): Only receive routine health education, without receiving individualized temperature health risk warning through the application

INTERVENTIONS:
Other: Temperature health risk early warning — Receive individualized temperature health risk warning through the application
  Arms: Temperature health risk early warning

SUMMARY:
This study applied an application to provide early warnings and advice for stroke patients and explored the impact of this intervention on reducing the risk of stroke recurrence

DETAILED DESCRIPTION:
This study applied an application that provides individualized environmental temperature-related health risk warnings and recommendations to stroke patients, enabling them to promptly understand their risk levels and take corresponding protective measures. And explore the effect of this actual intervention on reducing the risk of stroke recurrence after one year, as well as changes in other health-related indicators.

ELIGIBILITY:
Inclusion Criteria:

* Aged 40 to 80, with no gender restrictions;

  * Acute ischemic stroke inpatients within 2 weeks of onset, where the onset time is the time when stroke symptoms appear or the last known normal time of the patient (when it is an onset during sleep or the symptom onset time cannot be accurately obtained due to aphasia, impaired consciousness, etc.);

    * Confirmed diagnosis of ischemic stroke by CT or MRI of the brain within 2 weeks after symptom onset;

      * Local residents (residing for ≥6 months); ⑤ Patients who voluntarily participate in the study, have high compliance, and can sign the informed consent form;

        * Patients who own a smartphone or other smart devices.

Exclusion Criteria:

* Patients diagnosed with other cerebrovascular diseases (hemorrhagic stroke, transient ischemic attack, cerebral venous sinus thrombosis, etc.) or non-cerebrovascular diseases;

  * Known pregnant or lactating women, or those who tested positive on a pregnancy test before cluster randomization;

    * Patients with other conditions that may affect participation in the trial (e.g., refractory hypertension, severe aphasia, etc.);

      * Patients undergoing psychiatric/psychological treatment that may contaminate the results; ⑤ Patients with a life expectancy of less than one year (e.g., coexisting malignant tumors, severe cardiopulmonary diseases, etc.); ⑥ Patients already participating in other interventional clinical studies that may influence the outcome assessment; ⑦ Patients for whom the investigator deems unsuitable for participation in this study or who may pose significant risks to the patients (e.g., cognitive impairment preventing understanding and/or compliance with the study procedures and/or follow-up).

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5092 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
1-year recurrence rate of stroke | Intervention at the 1-year

SECONDARY OUTCOMES:
3-month, 6-month, 9-month recurrence rate of stroke | Intervention at 3-month, 6-month, 9-month
Blood pressure | Baseline; Intervention at 3-month, 6-month, 9-month and 1-year
  Systolic and diastolic blood pressure will be measured using a standard automated sphygmomanometer
Electrocardiogram (ECG) parameters | Baseline; Intervention at 3-month, 6-month, 9-month and 1-year
  Electrocardiogram (ECG) will be performed to assess cardiac electrical activity. Specific parameters will be analyzed, such as heart rate (beats per minute (bpm)), QT interval (milliseconds (ms)), PR interval (milliseconds (ms)), QRS duration (milliseconds (ms))
Environmental temperature health risk perception assessment questionnaire | Baseline; Intervention at 3-month, 6-month, 9-month and 1-year
  It is used to assess patients' understanding and concern about health hazards related to temperature. The lower the score, the less they understand or are concerned about it
System usability scale score | Intervention at 3-month, 6-month, 9-month and 1-year
  It is used to understand the subjects' satisfaction and usability evaluation of the intelligent program. The higher the score, the better the evaluation
Lipid Profile (Total Cholesterol, LDL-C, HDL-C, and Triglycerides) | Baseline; Intervention at 3-month, 6-month, 9-month and 1-year
  Plasma lipid levels will be measured using standard laboratory assays, including total cholesterol (TC), low-density lipoprotein cholesterol (LDL-C), high-density lipoprotein cholesterol (HDL-C), and triglycerides (TG).
Fasting blood glucose | Baseline; Intervention at 3-month, 6-month, 9-month and 1-year
  Fasting plasma glucose levels will be measured to assess glycemic control.
Coagulation parameters (Prothrombin Time, aPTT, INR, Fibrinogen, Platelet Count and D-dimer) | Baseline; Intervention at 3-month, 6-month, 9-month and 1-year
  Coagulation status will be assessed using standard coagulation tests, including prothrombin time (PT), activated partial thromboplastin time (aPTT), international normalized ratio (INR), fibrinogen level, platelet count and D-dimer.
C-reactive protein | Baseline; Intervention at 3-month, 6-month, 9-month and 1-year
  Blood samples will be analyzed using immunoassay techniques on automated analyzers
Modified rankin scale score | Baseline; Intervention at 3-month, 6-month, 9-month and 1-year
  The functional recovery of patients was evaluated using the modified rankin scale. The higher the score, the more serious it is
NIH stroke scale score | Baseline
  The neurological deficits on the NIHSS scale indicate that the higher the score, the more severe the stroke
European five-dimensional five-level health scale score | Baseline; Intervention at 3-month, 6-month, 9-month and 1-year
  It is used to assess an individual's health-related quality of life, consisting of two parts: a questionnaire and a visual analog scale (VAS). The questionnaire includes five dimensions, where higher scores indicate worse health status. The visual analog scale asks respondents to rate their overall health on a 0-100 scale, with higher scores reflecting better self-rated health status.
Minimum mental state examination | Baseline; Intervention at 6-month and 1-year
  It is used to screen patients' cognitive conditions. The lower the score, the worse the cognition
Social support rate scale score | Baseline; Intervention at 3-month, 6-month, 9-month and 1-year
  It is used to understand the support that patients receive in society, and the higher the score, the more support they receive
Depression anxiety stress scales - 21 score | Baseline; Intervention at 3-month, 6-month, 9-month and 1-year
  It is used to understand the patient's emotional state. The higher the score, the worse the mood

OTHER OUTCOMES:
Incidence of adverse cerebrovascular events | Intervention at the 1-year

CONTACTS AND LOCATIONS:
Overall Officials: Junwei Hao, Study Chair — Xuanwu Hospital, Beijing

IPD SHARING:
Plan to Share IPD: No